CLINICAL TRIAL: NCT03076411
Title: A Non-interventional, Observational Study With a Fixed Combination of Pepsin and Amino Acid Hydrochloride in Patients With Functional Dyspepsia
Brief Title: Pepsin in Patients With Functional Dyspepsia
Status: Completed | Type: Observational
Sponsor: Nordmark Arzneimittel GmbH & Co. KG (Industry)
Collaborators: ClinSupport GmbH (Industry); MWI Medizinisches Wirtschaftsinstitut GmbH (Unknown); das forschungsdock (Unknown)
Responsible Party: Sponsor
Other Study IDs: NM-Efo-401
Record Dates: First submitted 2016-10-19; First posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Functional Gastrointestinal Disorders; Abdominal Pain; Dyspepsia; Nausea; Vomiting; Flatulence
Keywords: Dyspepsia; Observational trial; Enzyme therapy; Pepsin
MeSH Terms: conditions — Gastrointestinal Diseases; Abdominal Pain; Dyspepsia; Nausea; Vomiting; Flatulence | interventions — Pepsin A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pepsin
  Other Names: amino acid hydrochloride

SUMMARY:
This non-interventional, observational study investigates the course of symptoms in patients with functional dyspepsia under treatment with a fixed combination of pepsin and amino acid hydrochloride over a period of approximately 6 weeks. The change of the Gastrointestinal Symptom Score (GIS©) was the primary parameter for the assessment of efficacy and was performed at baseline, after 3 and 6 weeks of treatment respectively. Safety measures included recording of AEs and physical examination as well as measurement of vital signs. The aim was to observe 100 patients during the course of this non-interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspepsia
* Women and men aged between 18 and 75

Exclusion Criteria:

- Unwilling to consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented with acute and chronic gastrointestinal symptoms, it was decided on the basis of their history, previous findings (diagnostic endoscopy and imaging, if available) and findings on physical examination whether they could participate in the postmarketing surveillance.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2013-12-19 (Actual); Study Completion 2015-06-16 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Score (GIS) | 6 weeks
  This is a third party assessment form.

SECONDARY OUTCOMES:
Tolerability assessed by Adverse Events | 6 weeks
  Adverse Events
Subjective assessment of efficacy (4 point Likert scale) | 6 weeks
  Patient overall assessment (very good, good, moderate, no effect)
Subjective assessment of feasibility of use (4 point Likert scale) | 6 weeks
  Patient overall assessment (very good, good, moderate, no effect)
Symptomatology | 6 weeks
  Nepean Dyspepsia Index (NDI) modified

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Forssmann, MD, Study Director — Nordmark Arzneimittel GmbH & Co. KG
Locations (1):
- Immanuel Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forssmann K, Meier L, Uehleke B, Breuer C, Stange R. A non-interventional, observational study of a fixed combination of pepsin and amino acid hydrochloride in patients with functional dyspepsia. BMC Gastroenterol. 2017 Nov 25;17(1):123. doi: 10.1186/s12876-017-0675-9. PMID 29178842